CLINICAL TRIAL: NCT04900376
Title: Evaluation of Covid-19 Vaccination in Elderly Subjects in Retirement Home (EHPAD) and Long-term Care Units (USLD) in Ile-de-France
Acronym: COGEVAX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A00007-34
Record Dates: First submitted 2021-05-22; First posted 2021-05-25 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Reside Either in Retirement Home or Long-term Care Units
Keywords: Retirement Home (EHPAD); Long-term Care Units (USLD); Coronavirus; Vaccination
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- vaccinated group
- unvaccinated group

SUMMARY:
The main objective of this non-interventional, multi-center study is to compare the incidence of serious health events (death, unscheduled hospitalizations) in subjects vaccinated against Coronavirus with that of unvaccinated subjects, in Retirement Home (EHPAD) and Long-term Care Units (USLD) in Ile-De-France during the same observation period 12-months minimun and up to18 months according vaccinal schedule.

The primary outcome will be the incidence of serious health events (death and unscheduled hospitalizations) in subjects vaccinated against Coronavirus compared to that of unvaccinated subjects.

DETAILED DESCRIPTION:
This multicenter study is a parallel cohort to the first phase of the vaccination campaign against Coronavirus, in particular for elderly subjects in institutions. All subjects who will not oppose the study will be included and this date will correspond to Day 0.

D0 will correspond to the date of the first vaccine injection for subjects in the vaccine group.

The subjects included will be followed up on D21, D90, M6, 12 months (M12) and up to 18 months in the case of 3rd vaccinal injection

The following data will be collected at inclusion and during follow-up:

* Age, weight, sex, level of autonomy
* Chronic diseases
* Any hospitalizations
* Possible symptoms after vaccination for subjects who choose to be vaccinated
* The fate of the subjects and the evaluation of the immune response
* Hospitalizations and vital status of subjects

Serology data prescribed by doctors as part of routine care will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Subject in Retirement Home (EHPAD) or Long-term Care Units (USLD) during the anti-Coronavivus vaccination period.
* Subject not opposing the study or whose legal representative does not oppose the study.

Exclusion Criteria:

* Subject not affiliated to a social security scheme.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Retirement Home (EHPAD) residents and Long-term Care Units (USLD) patients vaccinated or not against Coronavivus.
Sampling Method: Non-Probability Sample
Enrollment: 4100 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of the incidence of serious events in subjects vaccinated against CORONAVIRUS compared to those not vaccinated using their number, percentage and 95% confidence interval and methods of survival analysis Kaplan Meier and Cox model | 12 months or 18 months in the case of the 3rd vaccinal injection

SECONDARY OUTCOMES:
Assessment of the incidence of geriatric syndromes using their number, percentage and 95% confidence interval and survival analysis methods: Kaplan Meier and Cox model | 3 months
Evaluating the Incidence of Organ Decompensations according Their Number, Percentage, and 95% Confidence Interval and Survival Analysis Methods: Kaplan Meier and Cox Model | 6 months
Assessment of the incidence of serious and non-serious side effects using their number, percentage and 95% confidence interval and survival analysis methods: Kaplan Meier and Cox model. Kaplan Meier and Cox model | 3 months
Comparison of the incidence of symptomatic and severe coronavirus in vaccinated and unvaccinated subjects using their number, percentage and 95% confidence interval and survival analysis methods: Kaplan Meier and Cox Model. Kaplan Meier and Cox model | 3 months

OTHER OUTCOMES:
Carrying out adjustment analyzes by multivariate logistic regressions on confounding factors | 3 months
Performing propensity score analyzes to balance the vaccinated and unvaccinated groups | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Hanon, MD PhD, Study Chair — Geriatric Department, Broca hospital
Locations (1):
- Geriatric Department, Broca Hospital, Paris, IIe-de-France, France